CLINICAL TRIAL: NCT04776655
Title: Phase III Study in mCRC Patients With RAS/BRAF Wild Type Tissue and RAS Mutated in LIquid BIopsy to Compare in First-line Therapy FOLFIRI Plus CetuxiMAb or BevacizumaB (LIBImAb Study)
Brief Title: Study in mCRC Patients RAS/BRAF wt Tissue and RAS Mutated LIquid BIopsy to Compare FOLFIRI Plus CetuxiMAb or BevacizumaB
Acronym: LIBImAb
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Collaborators: Istituto Di Ricerche Farmacologiche Mario Negri (Other); Istituto Nazionale Tumori IRCCS - Fondazione G. Pascale (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-005078-82
Record Dates: First submitted 2021-02-23; First posted 2021-03-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer; Metastatic Colorectal Cancer; RAS Mutation
Keywords: mCRC; liquid biopsy; RAS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Cetuximab; Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Intervention Model Description: Phase III, randomized, open-label, comparative, multi-centre study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bevacizumab in combination with FOLFIRI chemotherapy (Experimental): Bevacizumab will be administrered at a dose of 5 mg/kg iv every 2 weeks. The first dose of Bevacizumab will be administered over 90 minutes. Then, if the first infusion is well tolerated without infusion-related reaction, the second dose will be administered over 60 minutes. Then, if the second dose is also well tolerated without an infusion reaction, all subsequent doses will be administered over 30 minutes.
  Dosage form: Intravenous use All treatments will continue until disease progression, death, unacceptable toxicity, clinical decision or consent withdrawn.
  Interventions: Drug: Bevacizumab; Drug: 5-FU; Drug: Irinotecan; Drug: Calcium levofolinate
- Cetuximab in combination with FOLFIRI chemotherapy (Active Comparator): Cetuximab will be administered at a dose of 500 mg/m² iv every 2 week (14 days/cycle) Dosage form: Intravenous use All treatments will continue until disease progression, death, unacceptable toxicity, clinical decision or consent withdrawn.
  Interventions: Drug: Cetuximab; Drug: 5-FU; Drug: Irinotecan; Drug: Calcium levofolinate

INTERVENTIONS:
Drug: Bevacizumab — This is the treatment assigned to experimental arm:
  All treatments will continue until disease progression, death, unacceptable toxicity, clinical decision or consent withdrawn.
  Other Names: Avastin
  Arms: Bevacizumab in combination with FOLFIRI chemotherapy
Drug: Cetuximab — This is the treatment assigned to control arm:
  All treatments will continue until disease progression, death, unacceptable toxicity, clinical decision or consent withdrawn.
  Other Names: Erbitux
  Arms: Cetuximab in combination with FOLFIRI chemotherapy
Drug: 5-FU — FOLFIRI regimen: This is the treatment assigned to control and to experimental arms:
  All treatments will continue until disease progression, death, unacceptable toxicity, clinical decision or consent withdrawn.
  Other Names: 5 Fluorouracil
Drug: Irinotecan — FOLFIRI regimen: This is the treatment assigned to control and to experimental arms:
  All treatments will continue until disease progression, death, unacceptable toxicity, clinical decision or consent withdrawn.
  Other Names: Irinotecano
Drug: Calcium levofolinate — FOLFIRI regimen: This is the treatment assigned to control and to experimental arms:
  All treatments will continue until disease progression, death, unacceptable toxicity, clinical decision or consent withdrawn.
  Other Names: Levofolinic acid

SUMMARY:
This study is a prospective, randomized phase III, to evaluate if in patients with mCRC RAS/BRAF wild type on tumor tissue and RAS mutations on liquid biopsy, treating in first line with antibody anti-VEGF (bevacizumab) plus chemotherapy (FOLFIRI) is superior in terms of PFS compared to standard treatment with antibody anti-EGFR (cetuximab) plus FOLFIRI, and then in patients RAS/BRAF wild type on tumor tissue who develop RAS mutations on liquid biopsy after the beginning of the first line treatment with cetuximab plus FOLFIRI, in the absence of a clinical or radiological progression disease, to anticipate a change of treatment with bevacizumab plus FOLFIRI further impacts on the PFS.

DETAILED DESCRIPTION:
In this prospective, randomized phase III study, first of all we aim to evaluate if in patients with mCRC RAS/BRAF wild type on tumor tissue and RAS mutations on liquid biopsy, treating in first line with antibody anti-VEGF (bevacizumab) plus chemotherapy (FOLFIRI) is superior in terms of PFS compared to standard treatment with antibody anti-EGFR (cetuximab) plus FOLFIRI, and then in patients RAS/BRAF wild type on tumor tissue who develop RAS mutations on liquid biopsy after the beginning of the first line treatment with cetuximab plus FOLFIRI, in the absence of a clinical or radiological progression disease, to anticipate a change of treatment with bevacizumab plus FOLFIRI further impacts on the PFS.

Patients RAS mut at first liquid biopsy will be randomized with a 1:1 ratio, to receive FOLFIRI plus cetuximab or FOLFIRI plus bevacizumab.

Patients with RAS wt at first biopsy will be treated with FOLFIRI plus cetuximab up to 8 cycles outside the protocol. Patients not progressed after 4 months (8 cycles of treatment) will undergo to a second liquid biopsy. In case of mutation of RAS, the patients will be randomized with a 1:1 ratio to continue cetuximab or to switch to bevacizumab.

The treatment will continue until disease progression, unacceptable toxicity, withdrawal of consent, other conditions compromise subject safety or patient refusal.

Plasma samples will be analyzed for mutations of KRAS, NRAS and in BRAF V600 using the Idylla system (Biocartis). Samples will be retrospectively analysed by next generation sequencing using the Oncomine Pan-Cancer Cell-free Assay, which assesses genetic alterations in 52 driver genes, in order to evaluate the possible correlation of tumor heterogeneity with patients' outcome.

With this study we could identify the best monoclonal antibody treatment in mCRC RAS/BRAF wild type on tumor tissue and RAS mutated on liquid biopsy and if liquid biopsy can be used in clinical practice as an integrated analysis to mutational tissue evaluation, to identify RAS mutations not detected on tissue.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent;
2. Male or female > 18 years of age;
3. Histologically confirmed diagnosis of colorectal adenocarcinoma RAS/BRAF wild type (analysed either on primary and/or related metastasis);
4. Initially unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease;
5. Patient with left colorectal cancer;
6. Patients suitable for first line chemotherapy;
7. Life expectancy > 3 months;
8. At least one site of measurable disease per RECIST criteria ver. 1.1;
9. ECOG Performance status = 2;
10. Adequate bone marrow, liver and renal function assessed before starting study treatment;
11. If DPD status is known it must be wild type. No restrictions are applied if DPD status in unknown;
12. Women of childbearing potential must have a negative blood pregnancy test within 24 hr prior to the start of study treatment. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 months, are surgically sterile, or are sexually inactive.
13. Subjects and their partners must be willing to avoid pregnancy during the trial and until 5 months for WOCBP (Women of Childbearing Potential) and 7 months for male subjects with female partners of WOCBP after the last trial treatment. Male subjects with female partners of childbearing potential and female subjects of childbearing potential must, therefore, be willing to use adequate contraception as approved by the investigator (barriers contraceptive measure or oral contraception).

Exclusion Criteria:

1. Previous chemotherapy treatment, with the exception of patient treated in adjuvant setting completed at least 6 months before the randomization;
2. Any contraindication to the use of Cetuximab, Bevacizumab, Irinotecan, 5FU or folinic acid;
3. Radiotherapy to any site within 4 weeks before the randomization;
4. Serious, non-healing wound, ulcer, or bone fracture;
5. Evidence of bleeding diathesis or coagulopathy;
6. Uncontrolled hypertension and prior history of hypertensive crisis or hypertensive encephalopathy;
7. Additional malignancy in the last 5 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy;
8. Active and untreated brain (CNS) metastases and/or carcinomatous meningitis;
9. Active infection requiring systemic therapy or active disseminated intravascular coagulation;
10. History of Human Immunodeficiency Virus (HIV) (HIV 1/2 antobodies);
11. Any positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection;
12. Chronic, daily treatment with high-dose aspirin (>325 mg/day);
13. Any previous venous thromboembolism > NCI CTCAE Grade 3;
14. History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to the first study treatment. History of acute or subacute intestinal occlusion or chronic inflammatory bowel disease or chronic diarrhoea;
15. Current, recent (within 10 days prior to study treatment start) or ongoing treatment with anticoagulants for therapeutic purposes;
16. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study;
17. History of any severe hypersensitivity reactions to any monoclonal antibody;
18. A significant concomitant disease which, in the investigating physician's opinion, rules out the patient's participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2025-05-04 (Actual); Study Completion 2026-05-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) in patients with RASmut at liquid biopsy and RASwt on tissue. | From the date of randomization to the date of first progression or death for any cause, whichever occurs first, assessed up to 36 months
  The primary objective of the study is to assess whether the combination of bevacizumab plus chemotherapy is superior to cetuximab plus chemotherapy in terms of progression free survival (PFS) in patients with RASmut at liquid biopsy and RASwt on tissue.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 36 months
  Overall survival (OS) defined as the time from start of treatment to the date of death for any cause or, for living patients, the date of last contact.
Objective response rate (ORR) | up to 36 months
  Objective Response Rate (ORR), defined as the percentage of patients with a complete (CR) or partial response (PR) as best response during treatment as determined by RECIST 1.1.
Prevalence of RAS mutation | up to 36 months
  Percentage of RAS mut patients on the total of patients who undergone to liquid biopsy at the first and second evaluations.
Patients Safety | up to 36 months
  The maximum toxicity grade experienced by each patient, for each toxicity, according to NCI-CTCAE v. 5.0; the number of patients experiencing grade 3-4 toxicity for each toxicity; type, frequency and nature of SAEs; patients with at least a SAE; patients with at least a SADR; patients with at least a SUSAR.
Compliance | up to 36 months
  The compliance to treatment will be described presenting number of administered cycles; frequency and reasons for drug discontinuation and treatment modifications.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Gervasi, Study Chair — AUSL IRCCS Reggio Emilia; Irene De Simone, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (4):
- Italy (4):
  - Ospedale San Salvatore, Coppito, L'Aquila
  - Ospedale Civile di Guastalla, Guastalla, Reggio Emilia
  - AUSL/IRCCS di Reggio Emilia, Reggio Emilia, Reggio Emilia
  - Azienda ULSS 3 Serenissima, Mirano, VE

IPD SHARING:
Plan to Share IPD: No